CLINICAL TRIAL: NCT03420690
Title: Study of the Impact of Art Therapy in Palliative Care on the Relationship Between Patients and Their Families
Acronym: ATREL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0626
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family of patient
  Interventions: Other: satisfaction questionnaire after art therapy session

INTERVENTIONS:
Other: satisfaction questionnaire after art therapy session — After the administration of art therapy sessions (>1) and the death of patients (> 1 month), the intervention consists in submitting to families of patients a satisfaction questionnaire intended to evaluate the impact of art therapy session and in particular about their relationships.

SUMMARY:
Negative symptoms in cancer in palliative care, such as pain, can lead to a withdrawal that can lead to a form of social exclusion. Maintaining pre-illness relationships is often difficult for the patient, especially since he is often not available to relationships.

Art therapy defined as the exploitation of artistic potential in a therapeutic and humanitarian aim can contribute to the reduction of symptoms, to adaptation and to well-being. A recent review shows that positive affective states and meaningful social connections are important factors contributing to more effective adaptation to pain. Study hypothesis is that art therapy could play on these two factors.

The objective of the qualitative study is to measure, using a questionnaire, the indirect impact of art therapy sessions on parents, during support and after death, from a relational and emotional point of view.

ELIGIBILITY:
Inclusion Criteria:

Any major person who has accompanied a patient to the palliative care unit of the Lyon-Sud hospital

* Man or woman ;
* 18 years old or older;
* Death of the accompanied patient> 1 month;
* Number of art therapy session of the accompanied patient > 1;
* Having agreed to participate in the study;
* Not subject to a legal protection measure.

Exclusion Criteria:

* Nobody without the physical or mental abilities to respond to the questionnaire ;
* No one reading or speaking French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Close to a patient who died more than 1 month old and who benefited from more than one art therapy session in the palliative care unit.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-06-24 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction with art therapy | 6 month
  The primary endpoint is the item of overall satisfaction with art therapy session in 3 groups (VAS scale between 0 and 3, between 3 and 7 and between 7 and 10)

CONTACTS AND LOCATIONS:
Overall Officials: Marilène FILBET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France